CLINICAL TRIAL: NCT01849666
Title: A PHASE I, OPEN-LABEL, MULTICENTER, RANDOMINZED, PARALELL STUDY TO INVESTIGATE THE EFFECT OF VEMURAFENIB ON THE PHARMACOKINETICS OF A SINGLE ORAL DOSE OF PHENPROCOUMON IN PATIENTS WITH BRAFV600 MUTATION-POSITIVE METASTATIC MALIGNANCY
Brief Title: A Study of the Effect of Vemurafenib on the Pharmacokinetics of Phenprocoumon in Patients With BRAFV600 Mutation-Positive Metastatic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GO28398; 2012-003707-35 (EudraCT Number)
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Malignant Melanoma, Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Phenprocoumon; Vemurafenib

ARMS (2):
- A: phenprocoumon single dose (Active Comparator)
  Interventions: Drug: phenprocoumon
- B: vemurafenib + phenprocoumon single dose (Experimental)
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: phenprocoumon — 6 mg oral single dose
  Arms: A: phenprocoumon single dose
Drug: vemurafenib — 960 mg bid orally
  Arms: B: vemurafenib + phenprocoumon single dose

SUMMARY:
This open-label, multicenter, parallel study will evaluate the effect of multiple doses of vemurafenib on the pharmacokinetics of a single dose of phenprocoumon in patients with BRAFV600 mutation-positive metastatic malignancies. Patients will be randomized to receive either treatment A: a single oral dose of phenprocoumon 6 mg on Day 1 (Eligible patients will have the option to continue treatment with vemurafenib as part of an extension study (NCT01739764).), or treatment B: vemurafenib 960 mg orally twice daily on Days 1-29 plus a single oral dose of phenprocoumon 6 mg on Day 22 (with the option to receive vemurafenib in the extension study after completion of pharmacokinetic assessments).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-70 years of age
* Patients with either unresectable Stage IIIc or IV BRAFV600 mutation-positive metastatic melanoma or other malignant BRAFV600 mutation-positive tumor type and who have no acceptable standard treatment options
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Full recovery from any major surgery or significant traumatic injury at least 14 days prior to the first dose of study treatment
* Adequate hematologic and end organ function
* Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use 2 effective methods of contraception as defined by protocol during the course of the study and for at least 6 months after completion of study treatment

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of Day 1
* Prior anti-cancer therapy within 28 days (6 weeks for nitrosureas or mitocyn C, or 14 days for hormonal therapy or kinase inhibitors) before the first dose of study treatment Day 1
* Palliative radiotherapy within 2 weeks prior to first dose of study treatment Day 1
* Experimental therapy within 4 weeks prior to first dose of study treatment Day 1
* History of clinically significant cardiac or pulmonary dysfunction, including current uncontrolled Grade >/=2 hypertension or unstable angina
* Current Grade >/=2 dyspnea or hypoxia or need for oxygen supplementation
* History of myocardial infarction within 6 months prior to first dose of study treatment
* Active central nervous system lesions (i.e. patients with radiographically unstable, symptomatic lesions)
* History of bleeding or coagulation disorders
* Allergy or hypersensitivity to vemurafenib or phenprocoumon formulations
* History of malabsorption or other condition that would interfere with the enteral absorption of study treatment
* History of clinically significant liver disease (including cirrhosis), current alcohol abuse, or active hepatitis B or hepatitis C virus infection
* Human immunodeficiency virus (HIV) infection requiring antiretroviral treatment, or AIDS-related illness
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single-dose phenprocoumon under conditions of vemurafenib steady-state exposure: Area under the concentration-time curve (AUC) | Pre-dose and up to 168 hours post-dose
Pharmacokinetics of single-dose phenprocoumon under conditions of vemurafenib steady-state exposure: Maximum plasma concentration (Cmax) | Pre-dose and up to 168 hours post-dose
Pharmacokinetics of single-dose phenprocoumon under conditions of vemurafenib steady-state exposure: Time to maximum plasma concentration (Tmax) | Pre-dose and up to 168 hours post-dose
Pharmacokinetics of single-dose phenprocoumon under conditions of vemurafenib steady-state exposure: Terminal half-life (t1/2) | Pre-dose and up to 168 hours post-dose
Pharmacokinetics of single-dose phenprocoumon under conditions of vemurafenib steady-state exposure: Apparent clearance (CL/F) | Pre-dose and up to 168 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence, nature and severity of adverse events (AEs) and serious AEs, graded according to NCI CTCAE Version 4.0 | approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Belgium (4):
  - Brussels
  - Edegem
  - Ghent
  - Wilrijk
- Helsinki, Finland
- Germany (2):
  - Heidelberg
  - Mainz
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Utrecht
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Pamplona, Navarre